CLINICAL TRIAL: NCT07183163
Title: Evaluating the Influence of Obesity on Peri-Implant Health Through Clinical and Biochemical Parameters
Brief Title: The Role of Obesity in Peri-Implant Health(ROPIPH)
Acronym: ROPIPH
Status: Completed | Type: Observational
Sponsor: Mine Keskin (Other)
Responsible Party: Sponsor-Investigator, Mine Keskin, Principal Investigator, Specialist in Periodontology, Recep Tayyip Erdogan University Faculty of Dentistry, Recep Tayyip Erdogan University
Organization: Recep Tayyip Erdogan University (Other)
Other Study IDs: E-40465587-050.01.04-432
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity &Amp; Overweight; Peri Implantitis; Dental Implant
Keywords: obesity; peri-implant health; dental implants; peri-implant sulcus fluid; inflamatory iomarkers (IL-1B, TNF-a, MMP-8)
MeSH Terms: conditions — Obesity; Overweight; Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PICF samples will be collected from implant sites using standardized paper strips. The samples will be analyzed for inflammatory biomarkers (IL-1beta, TNF-alfa, MMP-8) by ELISA. No DNA extraction will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- peri-implant healthy non-obese control group,: Clinically, the absence of signs of inflammation, bleeding and/or suppuration on probing, and any changes in the crestal bone levels other than bone remodeling were considered as peri-implant health. The presence of bleeding and/or suppuration on probing, a probing depth of 6 mm, and the presence of bone levels observed 3 mm apical to the most coronal part of the intraosseous part of the implant were considered as peri-implantitis. Participants with a BMI> 30 kg/m2 or waist circumference (WC): >100 cm in men and >90 cm in women were considered obese. According to their own statements, tobacco smokers, people who used smokeless tobacco products, those who used alcohol continuously, those who were pregnant or lactating, patients with systemic diseases such as acquired immune deficiency syndrome/HIV, kidney disorders, CVD, DM, and patients who had undergone any periodontal/periimplantitis treatment in the last 6 months were excluded from the study.
  Interventions: Other: Clinical and biochemical assessment
- periimplantitis non-obese group: Clinically, the absence of signs of inflammation, bleeding and/or suppuration on probing, and any changes in the crestal bone levels other than bone remodeling were considered as peri-implant health. The presence of bleeding and/or suppuration on probing, a probing depth of 6 mm, and the presence of bone levels observed 3 mm apical to the most coronal part of the intraosseous part of the implant were considered as peri-implantitis. Participants with a BMI> 30 kg/m2 or waist circumference (WC): >100 cm in men and >90 cm in women were considered obese. According to their own statements, tobacco smokers, people who used smokeless tobacco products, those who used alcohol continuously, those who were pregnant or lactating, patients with systemic diseases such as acquired immune deficiency syndrome/HIV, kidney disorders, CVD, DM, and patients who had undergone any periodontal/periimplantitis treatment in the last 6 months were excluded from the study.
  Interventions: Other: Clinical and biochemical assessment
- peri-implant healthy obese group: Clinically, the absence of signs of inflammation, bleeding and/or suppuration on probing, and any changes in the crestal bone levels other than bone remodeling were considered as peri-implant health. The presence of bleeding and/or suppuration on probing, a probing depth of 6 mm, and the presence of bone levels observed 3 mm apical to the most coronal part of the intraosseous part of the implant were considered as peri-implantitis. Participants with a BMI> 30 kg/m2 or waist circumference (WC): >100 cm in men and >90 cm in women were considered obese. According to their own statements, tobacco smokers, people who used smokeless tobacco products, those who used alcohol continuously, those who were pregnant or lactating, patients with systemic diseases such as acquired immune deficiency syndrome/HIV, kidney disorders, CVD, DM, and patients who had undergone any periodontal/periimplantitis treatment in the last 6 months were excluded from the study.
  Interventions: Other: Clinical and biochemical assessment
- periimplantitis obese group: Clinically, the absence of signs of inflammation, bleeding and/or suppuration on probing, and any changes in the crestal bone levels other than bone remodeling were considered as peri-implant health. The presence of bleeding and/or suppuration on probing, a probing depth of 6 mm, and the presence of bone levels observed 3 mm apical to the most coronal part of the intraosseous part of the implant were considered as peri-implantitis. Participants with a BMI> 30 kg/m2 or waist circumference (WC): >100 cm in men and >90 cm in women were considered obese. According to their own statements, tobacco smokers, people who used smokeless tobacco products, those who used alcohol continuously, those who were pregnant or lactating, patients with systemic diseases such as acquired immune deficiency syndrome/HIV, kidney disorders, CVD, DM, and patients who had undergone any periodontal/periimplantitis treatment in the last 6 months were excluded from the study.
  Interventions: Other: Clinical and biochemical assessment

INTERVENTIONS:
Other: Clinical and biochemical assessment — Assessment of peri-implant clinical parameters (probing depth, bleeding on probing, plaque index) and biochemical markers (IL-1β, TNF-α, MMP-8) in peri-implant crevicular fluid. No therapeutic or experimental intervention administered.

SUMMARY:
This clinical study aims to evaluate the influence of obesity on peri-implant health. Both clinical parameters and biochemical markers in peri-implant crevicular fluid(PICF) will be assessed. The study will include patients with dental implants who are classified as obese as well as a control group of non-obese participants. Clinical outcomes such as probing depth, plaque index, bleeding on probing, and peri-implant bone levels will be recorded. In addition, PICF samples will be analyzed for inflammatory biomarkers including interleukin-1 beta(IL-1beta), tumor necrosis factor-alpha(TNF-alfa), and matrix metalloproteinase-8(MMP-8). The results of this study may help to clarify the relationship between obesity and inflammatory responses in peri-implant tissues.

DETAILED DESCRIPTION:
This prospective clinical study investigates the role of obesity in peri-implant health by assessing both clinical and biochemical parameters. The study population will consist of systemically healthy individuals aged 18 years or older who have undergone dental implant treatment. Participants will be categorized into obese and non-obese groups according to body mass index (BMI) and waist circumference measurements. Clinical evaluations will include plaque index, bleeding on probing, probing depth, and radiographic assessment of peri-implant marginal bone loss. PICF will be collected from implant sites using standardized paper strips. The collected fluid will be analyzed for inflammatory biomarkers, including IL-1 beta, TNF-alfa, and MMP-8 using enzyme-linked immunosorbent assay (ELISA). The primary objective of the study is to determine whether obesity is associated with altered peri-implant clinical parameters and increased levels of inflammatory biomarkers. By correlating clinical and biochemical findings with obesity-related measures (BMI and waist circumference), this study aims to provide valuable insights into the potential impact of obesity on peri-implant tissue health and the risk of peri-implant diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with dental implants in function for at least 1 year.
* Patients diagnosed with peri-implantitis according to clinical and radiographic criteria.
* For control group: systemically healthy individuals with peri-implant health.
* Written informed consent obtained.

Exclusion Criteria:

* Patients with systemic diseases affecting periodontal/implant health (e.g., uncontrolled diabetes, HIV, cardiovascular disease, kidney disorders).
* Pregnant or lactating women.
* Current smokers or individuals using smokeless tobacco.
* Alcohol abuse.
* Use of antibiotics or anti-inflammatory drugs within the last 3 months.
* Patients who had received peri-implant treatment within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of systemically healthy adults aged 18-65 years with dental implants in function for at least 1 year. Participants will be categorized into obese and non-obese groups according to BMI and waist circumference measurements.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Levels of TNF-alfa in PICF | Baseline
  TNF-alfa concentration in PICF will be quantified using ELISA. Samples will be collected from four sites per implant (mesial, distal, buccal, lingual). Higher levels indicate increased inflammation.
Levels of IL-1 beta in PICF | Baseline
  IL-1beta concentration in PICF will be quantified using ELISA. Samples will be collected from four sites per implant (mesial, distal, buccal, lingual). Higher levels indicate increased inflammation.
Levels of MMP-8 in PICF | Baseline
  MMP-8 concentration in PICF will be quantified using ELISA. Samples will be collected from four sites per implant (mesial, distal, buccal, lingual). Higher levels indicate increased inflammation.

SECONDARY OUTCOMES:
Probing depth around dental implants | Baseline
  Probing depth will be measured at six sites per implant using a periodontal probe. The mean value per implant will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Department of Periodontology, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and institutional policy constraints. Only aggregated, de-identified summary results will be reported in the publication.